CLINICAL TRIAL: NCT05580224
Title: Anatomical Radiofrequency Ablation for Peripherally Located Small Hepatocellular Carcinoma Using Combined Energy Delivery Mode and Triple Cooled-Wet Electrodes
Brief Title: Anatomical Radiofrequency Ablation for Small Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2208-187-1355
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with hepatocellular carcinoma (equal or less than 3 cm) (Experimental): Under the guidance of multimodality-ultrasound (US) fusion image, one of the three electrodes was placed across the portal vein branch near the tumor, and the other two electrodes were placed around the tumor through the previously planned approach path. After placement of electrodes, the temperature is maintained at 90-100 degrees Celsius for about 6-30 minutes depending on the size of the tumor, using the combined energy transfer mode that sequentially adds the bipolar mode and/or the monopolar mode.
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Radiofrequency ablation — Radiofrequency ablation is performed for peripherally located small hepatocellular carcinoma using combined energy delivery mode and triple cooled-wet electrodes. One of three electrodes is placed across the 4th or 5th portal vein branches near the target tumor which enables anatomical ablation of tumor.

SUMMARY:
The aim of this study is to investigate therapeutic outcomes of anatomical radiofrequency ablation for peripherally located small hepatocellular carcinoma using combined energy delivery mode and triple cooled-wet electrodes.

ELIGIBILITY:
Inclusion Criteria:

* Child-Pugh class A or B7.
* Presence of chronic hepatitis B or liver cirrhosis.
* Patients with hepatocellular carcinomas diagnosed by histopathology or noninvasive imaging-based diagnosis according to the Korean Liver Cancer Association-National Cancer Center Korea guidelines.
* Patients with viable hepatocellular carcinoma after locoregional treatment diagnosed by the Liver Imaging Reporting and Data System.
* Tumor location is less than 5 cm from liver capsule.

Exclusion Criteria:

* The number of tumor is three or more.
* Tumor size is over 3 cm.
* Tumor location is over 5 cm from liver capsule.
* Child-Pugh class B8-9 or C.
* Presence of macrovascular invasion and/or distant metastasis.
* Platelet count < 50,000 mm3, or international normalized ratio > 1.5 (prothrombin time >1.5 × normal).

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2022-10-04 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Technical success | Immediately after radiofrequency ablation
  Technical success addresses whether the index tumor was treated according to a predefined protocol and entirely covered by the ablation zone.
Local tumor progression rate | 12 months after radiofrequency ablation
  Local tumor progression, defined as the appearance of tumor foci at the margin of the ablation zone after the attainment of treatment success.

SECONDARY OUTCOMES:
Complication after radiofrequency ablation | Immediately, 1 month, 3 months, 6 months, 9 months, and 12 months after radiofrequency ablation
  Post-radiofrequency ablation complications were defined as problems noted within 1 month after RFA as well as additional complications identified on follow-up imaging and judged to be likely caused by radiofrequency ablation.
Recurrence-free survival | 12 months after radiofrequency ablation
  Recurrence-free survival was defined as the interval between radiofrequency ablation and the date of any type of recurrence or the last follow-up date if there was no recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea